CLINICAL TRIAL: NCT04460404
Title: The Predictive Value of Alarm Symptoms in Patients With Function Constipation Based on Roman IV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 20200626
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Function Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle consultation — Collect relevant data of patients included in the study through outpatient consultation, telephone follow-up, questionnaire follow-up, etc., including:
  1. Basic information
  2. Digestive tract symptoms:
     A constipation-related symptoms B abnormal symptoms
  3. Fecal traits
  4. Lifestyle habits
  5. Others

SUMMARY:
Functional constipation is one of the five most common gastrointestinal diseases in outpatient visits. It is known that the global prevalence of chronic constipation is estimated to be 14%, and the prevalence of adults in my country is about 4.0% to 10.0%. It is generally believed that the diagnosis of functional constipation is based on a thorough history and physical examination. However, these standards are mainly used in clinical research and are not always strictly applicable to clinical practice. Therefore, in addition to the main symptoms, the medical history should include evidence of organic diseases (alarm symptoms). Rectal bleeding, anemia, weight loss, fever, family history of colon cancer and the age of onset over 50 years are considered as alarm symptoms of severe gastrointestinal diseases, but the value of alarm symptoms in distinguishing organic diseases from functional diseases is still not Ok, further research is still needed. In 2016, the Rome IV standard was updated and released, with some updates in the definition and diagnostic criteria for functional constipation. However, there are few studies on the clinical practice based on Rome IV. The advantages and disadvantages of adjusting the diagnostic criteria of Rome IV compared to Rome III in clinical application are still unclear. In order to evaluate the predictive value of the alarm symptoms of functional constipation based on Roman IV, we designed this cross-sectional study. It is used to evaluate the predictive value of alarm symptoms for functional constipation and organic bowel disease, as well as the predictive value of alarm symptoms of benign and malignant intestinal diseases related to functional constipation symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with constipation that meet the diagnostic criteria for functional constipation in Rome III or IV (specific conditions are as follows) (1) Must include two or more of the following:

   1. More than 25% of bowel movements feel laborious;
   2. Over 25% of the bowel movements are dry ball dung or hard dung; (Bristol Manure Character Scale Type 1-2)
   3. More than 25% of bowel movements have an inexhaustible feeling;
   4. More than 25% of bowel movements require manual assistance;
   5. More than 25% of bowel movements need to be assisted by manual techniques (such as assisting bowel movements with fingers and basin support);
   6. Less than 3 times per week (spontaneous defecation). (2) Dirty feces rarely occur when laxatives are not used. (3) Does not meet the diagnostic criteria for irritable bowel syndrome. (Symptoms appear at least 6 months before diagnosis, and meet the above (existence) diagnostic criteria within the past 3 months)
2. Age ≥18 years old;
3. From 2020.07 to 2020.12, visit the outpatient clinic of our hospital and perform colonoscopy;
4. Blood routine, fecal routine and fecal occult blood examination within 6 months.

Exclusion Criteria:

1. Inflammatory bowel disease, celiac disease and other organic intestinal diseases, history of metabolic diseases (abnormal thyroid function and diabetes, etc.);
2. Severe neurological, mental and psychological diseases, or those with severe organ dysfunction;
3. Abdominal surgery;
4. Patients during pregnancy, possible pregnancy and lactation;
5. Those who have a history of colonoscopy within the past 6 months, and those who have evaluated intestinal status;
6. Refuse to participate in this study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with constipation that meet the Rome IV diagnostic criteria are the subjects
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
the predictive value of alarm symptoms for functional constipation | 2020/12/31
  When a patient with constipation is accompanied by one or several alarm symptoms, the result of colonoscopy is confirmed as organic bowel disease
Predictive value of warning symptoms to malignant intestinal tumors | 2020/12/31
  When a patient with constipation is accompanied by one or more alarm symptoms, the result of colonoscopy is confirmed as malignant intestinal tumor

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No